CLINICAL TRIAL: NCT02141854
Title: A 12-Week, Double-Blind, Placebo-Controlled, Efficacy and Safety Study of Fluticasone Propionate Multidose Dry Powder Inhaler Compared With Fluticasone/Salmeterol Multidose Dry Powder Inhaler in Adolescent and Adult Patients With Persistent Asthma Symptomatic Despite Inhaled Corticosteroid Therapy
Brief Title: Efficacy and Safety Study of FP MDPI Compared With FS MDPI in Adolescent and Adult Patients With Persistent Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FSS-AS-30017; 2014-000923-25 (EudraCT Number)
Record Dates: First submitted 2014-05-09; First posted 2014-05-20 (Estimated); Results first posted 2017-04-12 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Fluticasone; Salmeterol Xinafoate; Albuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- FS MDPI 200 / 12.5 mcg (Experimental): Participants took 1 inhalation using a multidose dry powder inhaler (MDPI) twice a day of fluticasone propionate 200 mcg (for a total daily dose of 400 mcg) and salmeterol 12.5 mcg (for a total daily dose of 25 mcg) for 12 weeks.
  Interventions: Drug: FS MDPI; Drug: Albuterol/salmeterol HFA MDI
- FS MDPI 100 / 12.5 mcg (Experimental): Participants took 1 inhalation using a multidose dry powder inhaler (MDPI) twice a day of fluticasone propionate 100 mcg (for a total daily dose of 200 mcg) and salmeterol 12.5 mcg (for a total daily dose of 25 mcg) for 12 weeks.
  Interventions: Drug: FS MDPI; Drug: Albuterol/salmeterol HFA MDI
- Fp MDPI 200 mcg (Experimental): Participants took 1 inhalation using a multidose dry powder inhaler (MDPI) twice a day of fluticasone propionate (Fp) for a total daily dose of 400 mcg for 12 weeks.
  Interventions: Drug: Fp MDPI; Drug: Albuterol/salmeterol HFA MDI
- Fp MDPI 100 mcg (Experimental): Participants took 1 inhalation using a multidose dry powder inhaler (MDPI) twice a day of fluticasone propionate (Fp) for a total daily dose of 200 mcg for 12 weeks.
  Interventions: Drug: Fp MDPI; Drug: Albuterol/salmeterol HFA MDI
- Placebo MDPI (Placebo Comparator): Participants took 1 inhalation using a multidose dry powder inhaler (MDPI) twice a day of placebo for 12 weeks.
  Interventions: Drug: Placebo MDPI; Drug: Albuterol/salmeterol HFA MDI

INTERVENTIONS:
Drug: FS MDPI — FS MDPI is an inhalation-driven multidose dry powder inhaler (MDPI) containing fluticasone propionate and salmeterol xinafoate dispersed in a lactose monohydrate excipient and contained within a reservoir. A metered dose of drug is delivered to a dose cup via an air pulse activated when the cap is opened.
  During the treatment period, participants were randomized to either fluticasone propionate/salmeterol MDPI 200/12.5 mcg or fluticasone propionate/salmeterol MDPI 100/12.5 mcg twice a day for a total daily dose of 200/25 mcg or 400/25 mcg.
  Participants were instructed to rinse their mouth and expectorate (not swallow) after study drug administration.
  Other Names: fluticasone propionate; inhaled corticosteroid; salmeterol xinafoate; β2 adrenoceptor agonist
  Arms: FS MDPI 100 / 12.5 mcg; FS MDPI 200 / 12.5 mcg
Drug: Fp MDPI — Fp MDPI is an inhalation-driven multidose dry powder inhaler (MDPI) containing fluticasone propionate (Fp) dispersed in a lactose monohydrate excipient and contained within a reservoir. A metered dose of drug is delivered to a dose cup via an air pulse activated when the cap is opened.
  During the treatment period, participants were randomized to either 200 mcg or 100 mcg of Fp one inhalation twice a day for a total daily dose of 400 mcg or 200 mcg.
  Participants were instructed to rinse their mouth and expectorate (not swallow) after study drug administration.
  Other Names: fluticasone propionate; inhaled corticosteroid
  Arms: Fp MDPI 100 mcg; Fp MDPI 200 mcg
Drug: Placebo MDPI — The placebo multidose dry powder inhaler (MDPI) was identical to the devices used to deliver active drug, and indistinguishable from the active treatments. Patients took one inhalation twice a day (approximately 12 hours apart). Patients were instructed to rinse their mouth and expectorate (not swallow) after study drug administration.
  Other Names: inert powder
  Arms: Placebo MDPI
Drug: Albuterol/salmeterol HFA MDI — Albuterol/salmeterol hydrofluoroalkane (HFA) metered dose inhaler (MDI) was supplied to participants throughout the study to be used as needed as a rescue medication.
  Other Names: short-acting β2-adrenergic agonists

SUMMARY:
The primary objective of this study was to evaluate the efficacy of fluticasone propionate (Fp) multidose dry powder inhaler (MDPI) and fluticasone propionate/salmeterol xinafoate (FS) MDPI when administered over 12 weeks in patients 12 years of age and older with persistent asthma.

DETAILED DESCRIPTION:
Study drug and placebo were supplied in Teva multidose dry powder inhaler (MDPI) devices and provided for participants to use at home. Participants performed spirometry at every visit. Each participant was given a diary at each visit for use until the next visit. Rescue medication (albuterol/salbutamol) was dispensed at each visit, if needed, as determined by the investigational center personnel.

ELIGIBILITY:
Inclusion Criteria:

1. Best pre-bronchodilator forced expiratory volume in 1 second (FEV1) of 40 to 85% of their predicted normal value.
2. Current Asthma Therapy: Patients must have a short-acting β2-agonist (for rescue use) for a minimum of 8 weeks before the Screening Visit (SV) and a qualifying dose of an inhaled corticosteroid (ICS). The ICS may be either as ICS monotherapy or as an ICS/long-acting beta agonist (LABA) combination. The ICS component of the patient's asthma therapy should be stable for a minimum of 1 month before providing consent.
3. Reversibility of Disease: Patients must have at least 15% reversibility (all patients) and at least a 200 mL increase from baseline FEV1 (patients age 18 and older) within 30 minutes after 2 to 4 inhalations of albuterol/salbutamol at the SV. Note: Patients who do not qualify for the study due to failure to meet reversibility will be permitted to perform a retest once within 7 days.
4. Patients must provide written informed consent/assent.. For minor patients (ages 12 to 17 years, or as applicable per local regulations), the written ICF must be signed and dated by the parent/legal guardian and the written assent form must be signed and dated by the patient (if applicable). Note: Age requirements are as specified by local regulations.
5. Outpatient >= 12 years of age on the date of consent/assent. In countries where the local regulations permit enrollment of adult patients only, patients must be 18 years of age and older.
6. Asthma diagnosis: The patient has a diagnosis of asthma as defined by the National Institute of Health (NIH). The asthma diagnosis has been present for a minimum of 3 months and has been stable (defined as no exacerbations and no changes in asthma medication) for at least 30 days.
7. The patient is able to perform acceptable and repeatable spirometry.
8. The patient is able to perform peak expiratory flow (PEF) with a handheld peak flow meter.
9. The patient is able to use a metered dose inhaler (MDI) device without a spacer device and a multidose dry powder inhaler (MDPI) device.
10. The patient is able to withhold (as judged by the investigator) his or her regimen of ICS or study drug, and rescue medication for at least 6 hours before the screening visit (SV) and before all treatment visits.
11. The patient/parent/legal guardian/caregiver is capable of understanding the requirements, risks, and benefits of study participation, and, as judged by the investigator, capable of giving informed consent/assent and being compliant with all study requirements.
12. SABAs: All patients must be able to replace their current SABA with albuterol/salbutamol HFA MDI inhalation aerosol for the duration of the study.
13. Female patients may not be pregnant, breastfeeding, or attempting to become pregnant.

    * other criteria may apply, please contact the investigator for more information

Exclusion Criteria:

1. A history of a life-threatening asthma exacerbation (an asthma episode that required intubation and/or was associated with hypercapnia, respiratory arrest, or hypoxic seizures).
2. The patient is pregnant or lactating, or plans to become pregnant during the study period or for 30 days after the study.
3. The patient has participated as a randomized patient in any investigational drug study within 30 days of the SV.
4. The patient has previously participated as a randomized patient in a study of Fp MDPI or FS MDPI.
5. The patient has a known hypersensitivity to any corticosteroid, salmeterol, or any of the excipients in the study drug or rescue medication formulation (ie, lactose).
6. The patient has been treated with any known strong cytochrome P450 (CYP) 3A4 inhibitors (eg, azole antifungals, ritonavir, or clarithromycin) within 30 days before the SV.
7. The patient has been treated with any of the prohibited medications during the prescribed (per protocol) washout periods before the SV.
8. The patient currently smokes or has a smoking history of 10 pack years or more (a pack year is defined as smoking 1 pack of cigarettes/day for 1 year). The patient must not have used tobacco products within the past year (eg, cigarettes, cigars, chewing tobacco, or pipe tobacco).
9. The patient has a culture-documented or suspected bacterial or viral infection of the upper or lower respiratory tract, sinus, or middle ear that has not resolved at least 2 weeks before the SV.
10. The patient has a history of alcohol or drug abuse within 2 years preceding the SV.
11. The patient has had an asthma exacerbation requiring systemic corticosteroids within 30 days before the SV, or has had any hospitalization for asthma within 2 months before the SV.
12. Initiation or dose escalation of immunotherapy (administered by any route) is planned during the study period. However, patients on stable immunotherapy may be considered for inclusion.
13. The patient has used immunosuppressive medications within 4 weeks before the SV.
14. The patient is unable to tolerate or unwilling to comply with the appropriate washout periods and withholding of all applicable medications.
15. The patient has untreated oral candidiasis at the SV. Patients with clinical visual evidence of oral candidiasis who agree to receive treatment and comply with appropriate medical monitoring may enter the study.
16. The patient has a history of a positive test for human immunodeficiency virus (HIV), active hepatitis B virus, or hepatitis C infection.
17. The patient is either an employee or an immediate relative of an employee of the clinical investigational center.
18. A member of the patient's household is participating in the study at the same time. However, after the enrolled patient completes or discontinues participation in the study, another patient from the same household may be screened.
19. The patient has a disease/condition that in the medical judgment of the investigator would put the safety of the patient at risk through participation or that could affect the efficacy or safety analysis if the disease/condition worsened during the study.

    * other criteria may apply, please contact the investigator for more information

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 882 (Actual)
Dates: Start 2014-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (154):
- United States (85):
  - Teva Investigational Site 12429, Birmingham, Alabama
  - Teva Investigational Site 12599, Little Rock, Alaska
  - Teva Investigational Site 12609, Phoenix, Arizona
  - Teva Investigational Site 12445, Costa Mesa, California
  - Teva Investigational Site 12454, Encinitas, California
  - Teva Investigational Site 12456, Fresno, California
  - Teva Investigational Site 12461, Fullerton, California
  - Teva Investigational Site 12410, Huntington Beach, California
  - Teva Investigational Site 12452, Huntington Beach, California
  - Teva Investigational Site 12417, Long Beach, California
  - Teva Investigational Site 13017, Mission Viejo, California
  - Teva Investigational Site 12462, Rancho Mirage, California
  - Teva Investigational Site 12411, Rolling Hills Estates, California
  - Teva Investigational Site 13018, San Diego, California
  - Teva Investigational Site 12413, San Jose, California
  - Teva Investigational Site 12403, Stockton, California
  - Teva Investigational Site 12444, Upland, California
  - Teva Investigational Site 12999, Vista, California
  - Teva Investigational Site 12405, Centennial, Colorado
  - Teva Investigational Site 12419, Centennial, Colorado
  - Teva Investigational Site 13000, Colorado Springs, Colorado
  - Teva Investigational Site 12459, Waterbury, Connecticut
  - Teva Investigational Site 13004, Largo, Florida
  - Teva Investigational Site 12414, Miami, Florida
  - Teva Investigational Site 12437, Miami, Florida
  - Teva Investigational Site 12427, Orlando, Florida
  - Teva Investigational Site 12423, Ormond Beach, Florida
  - Teva Investigational Site 12604, Panama City, Florida
  - Teva Investigational Site 13316, Tamarac, Florida
  - Teva Investigational Site 12606, Winter Park, Florida
  - Teva Investigational Site 12435, Savannah, Georgia
  - Teva Investigational Site 13315, Eagle, Idaho
  - Teva Investigational Site 12439, River Forest, Illinois
  - Teva Investigational Site 12449, Shiloh, Illinois
  - Teva Investigational Site 12457, South Bend, Indiana
  - Teva Investigational Site 12446, Bangor, Maine
  - Teva Investigational Site 12602, Columbia, Maryland
  - Teva Investigational Site 12432, Fall River, Massachusetts
  - Teva Investigational Site 12441, North Dartmouth, Massachusetts
  - Teva Investigational Site 12466, North Dartmouth, Massachusetts
  - Teva Investigational Site 13001, Royal Oak, Michigan
  - Teva Investigational Site 12428, Ypsilanti, Michigan
  - Teva Investigational Site 13020, Minneapolis, Minnesota
  - Teva Investigational Site 12451, Columbia, Missouri
  - Teva Investigational Site 12421, Rolla, Missouri
  - Teva Investigational Site 12412, St Louis, Missouri
  - Teva Investigational Site 12453, St Louis, Missouri
  - Teva Investigational Site 12610, Missoula, Montana
  - Teva Investigational Site 13021, Las Vegas, Nevada
  - Teva Investigational Site 12409, Skillman, New Jersey
  - Teva Investigational Site 12464, Brooklyn, New York
  - Teva Investigational Site 12603, The Bronx, New York
  - Teva Investigational Site 12430, Charlotte, North Carolina
  - Teva Investigational Site 12407, Raleigh, North Carolina
  - Teva Investigational Site 12415, Canton, Ohio
  - Teva Investigational Site 12455, Cincinnati, Ohio
  - Teva Investigational Site 12463, Cincinnati, Ohio
  - Teva Investigational Site 12460, Middleburg Heights, Ohio
  - Teva Investigational Site 12426, Edmond, Oklahoma
  - Teva Investigational Site 13008, Oklahoma City, Oklahoma
  - Teva Investigational Site 12406, Medford, Oregon
  - Teva Investigational Site 12442, Portland, Oregon
  - Teva Investigational Site 12563, Normal Square, Pennsylvania
  - Teva Investigational Site 12443, Pittsburgh, Pennsylvania
  - Teva Investigational Site 12438, Upland, Pennsylvania
  - Teva Investigational Site 12408, Charleston, South Carolina
  - Teva Investigational Site 12431, Greenville, South Carolina
  - Teva Investigational Site 12465, Mt. Pleasant, South Carolina
  - Teva Investigational Site 12467, Mt. Pleasant, South Carolina
  - Teva Investigational Site 12420, Orangeburg, South Carolina
  - Teva Investigational Site 12433, Rock Hill, South Carolina
  - Teva Investigational Site 13003, Knoxville, Tennessee
  - Teva Investigational Site 12425, Arlington, Texas
  - Teva Investigational Site 12416, Dallas, Texas
  - Teva Investigational Site 12418, Dallas, Texas
  - Teva Investigational Site 12440, El Paso, Texas
  - Teva Investigational Site 12447, Killeen, Texas
  - Teva Investigational Site 13318, San Antonio, Texas
  - Teva Investigational Site 13002, Sugar Land, Texas
  - Teva Investigational Site 12424, Waco, Texas
  - Teva Investigational Site 12422, South Burlington, Vermont
  - Teva Investigational Site 12605, Richmond, Virginia
  - Teva Investigational Site 12436, Spokane, Washington
  - Teva Investigational Site 12564, Tacoma, Washington
  - Teva Investigational Site 12448, Greenfield, Wisconsin
- Canada (2):
  - Teva Investigational Site 11072, Toronto, Ontario
  - Teva Investigational Site 11075, Vancouver, Quebec
- Czechia (4):
  - Teva Investigational Site 54096, Jindřichův Hradec
  - Teva Investigational Site 54098, Prague
  - Teva Investigational Site 54095, Rokycany
  - Teva Investigational Site 54094, Strakonice
- Hungary (18):
  - Teva Investigational Site 51149, Budapest
  - Teva Investigational Site 51155, Budapest
  - Teva Investigational Site 51157, Budapest
  - Teva Investigational Site 51161, Budapest
  - Teva Investigational Site 51154, Debrecen
  - Teva Investigational Site 51152, Deszk
  - Teva Investigational Site 51170, Dombóvár
  - Teva Investigational Site 51158, Kiskunhalas
  - Teva Investigational Site 51153, Miskolc
  - Teva Investigational Site 51156, Mosdós
  - Teva Investigational Site 51150, Nyíregyháza
  - Teva Investigational Site 51151, Nyíregyháza
  - Teva Investigational Site 51148, Százhalombatta
  - Teva Investigational Site 51146, Szeged
  - Teva Investigational Site 51162, Szigetvár
  - Teva Investigational Site 51147, Szombathely
  - Teva Investigational Site 51176, Tatabánya
  - Teva Investigational Site 51177, Törökbálint
- Poland (23):
  - Teva Investigational Site 53199, Bialystok
  - Teva Investigational Site 53200, Bialystok
  - Teva Investigational Site 53202, Bialystok
  - Teva Investigational Site 53208, Bialystok
  - Teva Investigational Site 53210, Bydgoszcz
  - Teva Investigational Site 53227, Bydgoszcz
  - Teva Investigational Site 53225, Dębica
  - Teva Investigational Site 53203, Gdansk
  - Teva Investigational Site 53195, Krakow
  - Teva Investigational Site 53197, Krakow
  - Teva Investigational Site 53205, Krakow
  - Teva Investigational Site 53228, Lodz
  - Teva Investigational Site 53240, Lodz
  - Teva Investigational Site 53201, Lódz
  - Teva Investigational Site 53229, Lódz
  - Teva Investigational Site 53241, Lublin
  - Teva Investigational Site 53206, Poznan
  - Teva Investigational Site 53211, Poznan
  - Teva Investigational Site 53230, Strzelce Opolskie
  - Teva Investigational Site 53196, Tarnów
  - Teva Investigational Site 53222, Warsaw
  - Teva Investigational Site 53198, Wroclaw
  - Teva Investigational Site 53224, Wroclaw
- Russia (12):
  - Teva Investigational Site 50255, Chelyabinsk
  - Teva Investigational Site 50241, Kazan'
  - Teva Investigational Site 50250, Moscow
  - Teva Investigational Site 50252, Moscow
  - Teva Investigational Site 50242, Saint Petersburg
  - Teva Investigational Site 50245, Saint Petersburg
  - Teva Investigational Site 50246, Saint Petersburg
  - Teva Investigational Site 50254, Saratov
  - Teva Investigational Site 50244, Tomsk
  - Teva Investigational Site 50251, Voronezh
  - Teva Investigational Site 50275, Yaroslavl
  - Teva Investigational Site 50243, Yekaterinburg
- South Africa (6):
  - Teva Investigational Site 90011, Berea
  - Teva Investigational Site 90015, Bloemfontein
  - Teva Investigational Site 90012, Cape Town
  - Teva Investigational Site 90013, Centurion
  - Teva Investigational Site 90016, Middelburg
  - Teva Investigational Site 90014, Pretoria
- Teva Investigational Site 12404, Papillion, NE, Thailand
- Ukraine (3):
  - Teva Investigational Site 58133, Kharkiv
  - Teva Investigational Site 58135, Kharkiv
  - Teva Investigational Site 58132, Kyiv

REFERENCES:
- [Derived] Sher LD, Yiu G, Sakov A, Liu S, Caracta CF. Fluticasone propionate and fluticasone propionate/salmeterol multidose dry powder inhalers compared with placebo for persistent asthma. Allergy Asthma Proc. 2017 Sep 21;38(5):343-353. doi: 10.2500/aap.2017.38.4069. Epub 2017 Jun 21. PMID 28639542
- [Derived] Miller DS, Yiu G, Hellriegel ET, Steinfeld J. Dose-ranging study of salmeterol using a novel fluticasone propionate/salmeterol multidose dry powder inhaler in patients with persistent asthma. Allergy Asthma Proc. 2016 Jul;37(4):291-301. doi: 10.2500/aap.2016.37.3963. Epub 2016 May 27. PMID 27216137

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1661 patients with persistent asthma were screened and 882 patients enrolled. 154 patients were not randomized, most commonly (76 patients) because of not meeting randomization criteria.
Groups:
- Fluticasone Propionate 50 mcg BID: All enrolled participants used single-blind fluticasone propionate multidose dry powder inhaler twice a day for a total daily dose of 100 mcg during the Run-In Period (14-21 days).
- FS MDPI 200 / 12.5 mcg: Following randomization, participants in this treatment arm took 1 inhalation twice a day using a multidose dry powder inhaler (MDPI) of fluticasone propionate 200 mcg (for a total daily dose of 400 mcg) and salmeterol 12.5 mcg (for a total daily dose of 25 mcg) for 12 weeks.
  Albuterol/salmeterol HFA MDI: Albuterol/salmeterol hydrofluoroalkane (HFA) metered dose inhaler (MDI) was supplied to participants throughout the study to be used as needed as a rescue medication.
- FS MDPI 100 / 12.5 mcg: Following randomization, participants in this treatment arm took 1 inhalation using a multidose dry powder inhaler (MDPI) twice a day of fluticasone propionate 100 mcg (for a total daily dose of 200 mcg) and salmeterol 12.5 mcg (for a total daily dose of 25 mcg) for 12 weeks.
  Albuterol/salmeterol HFA MDI: Albuterol/salmeterol hydrofluoroalkane (HFA) metered dose inhaler (MDI) was supplied to participants throughout the study to be used as needed as a rescue medication.
- Fp MDPI 200 mcg: Following randomization, participants in this treatment arm took 1 inhalation using a multidose dry powder inhaler (MDPI) twice a day of fluticasone propionate (Fp) for a total daily dose of 400 mcg for 12 weeks.
  Albuterol/salmeterol HFA MDI: Albuterol/salmeterol hydrofluoroalkane (HFA) metered dose inhaler (MDI) was supplied to participants throughout the study to be used as needed as a rescue medication.
- Fp MDPI 100 mcg: Following randomization, participants in this treatment arm took 1 inhalation using a multidose dry powder inhaler (MDPI) twice a day of fluticasone propionate (Fp) for a total daily dose of 200 mcg for 12 weeks.
  Albuterol/salmeterol HFA MDI: Albuterol/salmeterol hydrofluoroalkane (HFA) metered dose inhaler (MDI) was supplied to participants throughout the study to be used as needed as a rescue medication.
- Placebo MDPI: Following randomization, participants in this treatment arm took 1 inhalation using a multidose dry powder inhaler (MDPI) twice a day of placebo for 12 weeks.
  Albuterol/salmeterol HFA MDI: Albuterol/salmeterol hydrofluoroalkane (HFA) metered dose inhaler (MDI) was supplied to participants throughout the study to be used as needed as a rescue medication.
Period: Run-In Period (Pre-assignment)
Arm/Group | Fluticasone Propionate 50 mcg BID | FS MDPI 200 / 12.5 mcg | FS MDPI 100 / 12.5 mcg | Fp MDPI 200 mcg | Fp MDPI 100 mcg | Placebo MDPI
Started | 882 | 0 | 0 | 0 | 0 | 0
Completed | 728 | 0 | 0 | 0 | 0 | 0
Not Completed | 154 | 0 | 0 | 0 | 0 | 0
Not completed — Inclusion criteria not met | 25 | 0 | 0 | 0 | 0 | 0
Not completed — Randomization criteria not met | 76 | 0 | 0 | 0 | 0 | 0
Not completed — Exclusion criteria met | 14 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 14 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 10 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 9 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 6 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period
Arm/Group | Fluticasone Propionate 50 mcg BID | FS MDPI 200 / 12.5 mcg | FS MDPI 100 / 12.5 mcg | Fp MDPI 200 mcg | Fp MDPI 100 mcg | Placebo MDPI
Started | 0 | 146 | 145 | 146 | 146 | 145
Intent to Treat Population | 0 | 146 | 145 | 146 | 146 | 145
Safety Population | 0 | 145 | 143 | 146 | 145 | 144
Full Analysis Set | 0 | 145 | 141 | 146 | 145 | 143
Completed | 0 | 136 | 136 | 135 | 136 | 107
Not Completed | 0 | 10 | 9 | 11 | 10 | 38
Not completed — Protocol Violation | 0 | 1 | 0 | 2 | 2 | 1
Not completed — Noncompliance | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1 | 1 | 7
Not completed — Pregnancy | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 1 | 2 | 0 | 1 | 2
Not completed — Adverse Event | 0 | 2 | 2 | 0 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 2 | 3 | 3 | 4 | 7
Not completed — Disease progression | 0 | 2 | 1 | 3 | 0 | 18
Not completed — Lost to Follow-up | 0 | 1 | 1 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | FS MDPI 200 / 12.5 mcg | FS MDPI 100 / 12.5 mcg | Fp MDPI 200 mcg | Fp MDPI 100 mcg | Placebo MDPI | Total
Number analyzed (Participants) | 146 | 145 | 146 | 146 | 145 | 728
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.7 (16.93) | 44.3 (14.88) | 44.4 (16.36) | 45.7 (15.64) | 44.5 (16.05) | 44.7 (15.95)
Age, Customized [Count of Participants; unit: Participants]
  Adolescents (12-17 years) | 12 | 8 | 10 | 9 | 6 | 45
  Adults (18-64 years) | 115 | 125 | 119 | 124 | 125 | 608
  Adults (65-84 years) | 19 | 12 | 17 | 13 | 14 | 75
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 79 | 88 | 94 | 91 | 439
  Male | 59 | 66 | 58 | 52 | 54 | 289
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 125 | 112 | 116 | 111 | 124 | 588
  Black or African American | 20 | 28 | 23 | 31 | 18 | 120
  Asian | 0 | 0 | 2 | 0 | 2 | 4
  American Indian or Alaskan Native | 0 | 0 | 2 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Other | 1 | 5 | 3 | 4 | 1 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 136 | 135 | 136 | 134 | 136 | 677
  Hispanic or Latino | 10 | 10 | 10 | 11 | 8 | 49
  Unknown | 0 | 0 | 0 | 1 | 1 | 2
History of Smoking [Count of Participants; unit: Participants]
  Prior Smoker | 20 | 28 | 21 | 28 | 23 | 120
  No tobacco use | 126 | 117 | 125 | 118 | 122 | 608
Previous Asthma Therapy [Count of Participants; unit: Participants]
  Inhaled corticosteroid | 73 | 67 | 63 | 58 | 68 | 329
  Inhaled corticosteroid/long-acting beta2-agonist | 73 | 78 | 83 | 88 | 77 | 399
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.4 (7.35) | 30.2 (7.60) | 29.9 (7.27) | 29.9 (7.62) | 29.3 (7.41) | 29.7 (7.44)
Forced Expiratory Volume in 1 second (FEV1) [Mean (Standard Deviation); unit: liters] — Population: Some participants were missing baseline values
  liters
    number analyzed (Participants) | 145 | 142 | 146 | 145 | 144 | 722
    (all) | 2.083 (0.6532) | 2.157 (0.6402) | 2.075 (0.5696) | 2.069 (0.6017) | 2.141 (0.6849) | 2.105 (0.6303)

OUTCOME MEASURES:

1. Primary Outcome: Standardized Baseline-Adjusted Forced Expiratory Volume in 1 Second (FEV1) Area Under the Effect Curve From Time Zero to 12 Hours PostDose (FEV1 AUEC0-12) at Week 12
Description: A subset of patients performed postdose serial spirometry. Data from these assessments were used to analyze the primary endpoint of baseline-adjusted FEV1 AUEC0-12h at week 12 using the trapezoidal rule based on actual time of measurement. It was standardized by dividing it by the number of hours between the start time of dose administration and the end time of the last nonmissing FEV1 measurement. The baseline FEV1 was the average of the 2 predose FEV1 measurements (30 and 10 minutes predose). If 1 of these was missing, the nonmissing value was used; if both were missing, baseline was treated as missing. Baseline-adjusted FEV1 was calculated as postdose FEV1 after subtracting the baseline FEV1 value.
Time Frame: Day 1 (predose, baseline), Week 12 and was performed at the following times relative to the administration of study drug (±5 minutes): 15 and 30 minutes and 1, 2, 3, 4, 6, 8, 10, and 12 hours
Population: A subset of patients who performed postdose serial spirometry at the baseline visit and week 12.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | FS MDPI 200 / 12.5 mcg | FS MDPI 100 / 12.5 mcg | Fp MDPI 200 mcg | Fp MDPI 100 mcg | Placebo MDPI
Number analyzed (Participants) | 68 | 58 | 61 | 64 | 61
liters | 0.446 (0.0463) | 0.442 (0.0496) | 0.267 (0.0466) | 0.260 (0.0463) | 0.121 (0.0472)
Statistical Analysis 1: Comparison: FS MDPI 200 / 12.5 mcg vs Fp MDPI 200 mcg; A fixed-sequence multiple testing procedure was used to control the overall Type I error rate at the 0.05 level (2-sided) for the primary endpoints analyses. Analyses appear in the defined sequence. This is the first in the sequence; Test type: Superiority or Other; p = 0.0009, ANCOVA — Fixed effects of treatment, sex, (pooled) center, previous therapy (ICS or ICS/LABA), and covariates of age and baseline FEV1; LSM difference = 0.179, 95% CI 2-sided [0.074 to 0.285]
Statistical Analysis 2: Comparison: FS MDPI 100 / 12.5 mcg vs Fp MDPI 100 mcg; A fixed-sequence multiple testing procedure was used to control the overall Type I error rate at the 0.05 level (2-sided) for the primary endpoints analyses. Analyses appear in the defined sequence. This is the second in the sequence; Test type: Superiority or Other; p = 0.0010, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LSM difference = 0.182, 95% CI 2-sided [0.074 to 0.291]
Statistical Analysis 3: Comparison: FS MDPI 200 / 12.5 mcg vs Placebo MDPI; A fixed-sequence multiple testing procedure was used to control the overall Type I error rate at the 0.05 level (2-sided) for the primary endpoints analyses. Analyses appear in the defined sequence. This is the third in the sequence; Test type: Superiority or Other; p = 0.0000, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LSM difference = 0.326, 95% CI 2-sided [0.221 to 0.431]
Statistical Analysis 4: Comparison: FS MDPI 100 / 12.5 mcg vs Placebo MDPI; A fixed-sequence multiple testing procedure was used to control the overall Type I error rate at the 0.05 level (2-sided) for the primary endpoints analyses. Analyses appear in the defined sequence. This is the fourth in the sequence; Test type: Superiority or Other; p = 0.0000, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LSM difference = 0.322, 95% CI 2-sided [0.212 to 0.432]

2. Primary Outcome: Change From Baseline in Morning Trough Forced Expiratory Volume in 1 Second (FEV1) at Week 12
Description: Trough FEV1 is a morning spirometry taken predose and pre-rescue bronchodilator. The baseline for predose FEV1 was defined as the average of the 30-minute and 10-minute predose measurements obtained at the randomization visit (Day 1).
Time Frame: Day 1 (predose, baseline), Week 12
Population: If the patient inadvertently administered asthma medication/study drug at home on the AM of the visit, or if the patient took rescue medication within 6 hours of testing, the visit was rescheduled.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | FS MDPI 200 / 12.5 mcg | FS MDPI 100 / 12.5 mcg | Fp MDPI 200 mcg | Fp MDPI 100 mcg | Placebo MDPI
Number analyzed (Participants) | 143 | 140 | 145 | 144 | 143
liters | 0.272 (0.0307) | 0.271 (0.0311) | 0.179 (0.0308) | 0.119 (0.0311) | -0.004 (0.0312)
Statistical Analysis 1: Comparison: FS MDPI 200 / 12.5 mcg vs Placebo MDPI; A fixed-sequence multiple testing procedure was used to control the overall Type I error rate at the 0.05 level (2-sided) for the primary endpoints analyses. Analyses appear in the defined sequence. This is the fifth in the sequence; Test type: Superiority or Other; p = 0.0000, ANCOVA — Effects due to baseline trough AM FEV1, sex, age, (pooled) center, previous therapy (ICS or ICS/LABA), and treatment; LSM difference = 0.276, 95% CI 2-sided [0.191 to 0.361]
Statistical Analysis 2: Comparison: FS MDPI 100 / 12.5 mcg vs Placebo MDPI; A fixed-sequence multiple testing procedure was used to control the overall Type I error rate at the 0.05 level (2-sided) for the primary endpoints analyses. Analyses appear in the defined sequence. This is the sixth in the sequence; Test type: Superiority or Other; p = 0.0000, ANCOVA — Effects due to baseline trough AM FEV1, sex, age, (pooled) center, previous therapy (ICS or ICS/LABA), and treatment; LSM difference = 0.274, 95% CI 2-sided [0.189 to 0.360]
Statistical Analysis 3: Comparison: Fp MDPI 200 mcg vs Placebo MDPI; A fixed-sequence multiple testing procedure was used to control the overall Type I error rate at the 0.05 level (2-sided) for the primary endpoints analyses. Analyses appear in the defined sequence. This is the seventh in the sequence; Test type: Superiority or Other; p = 0.0000, ANCOVA — Effects due to baseline trough AM FEV1, sex, age, (pooled) center, previous therapy (ICS or ICS/LABA), and treatment; LSM difference = 0.183, 95% CI 2-sided [0.098 to 0.268]
Statistical Analysis 4: Comparison: Fp MDPI 100 mcg vs Placebo MDPI; A fixed-sequence multiple testing procedure was used to control the overall Type I error rate at the 0.05 level (2-sided) for the primary endpoints analyses. Analyses appear in the defined sequence. This is the eighth in the sequence; Test type: Superiority or Other; p = 0.0047, ANCOVA — Effects due to baseline trough AM FEV1, sex, age, (pooled) center, previous therapy (ICS or ICS/LABA), and treatment; LSM difference = 0.123, 95% CI 2-sided [0.038 to 0.208]

3. Secondary Outcome: Change From Baseline in the Weekly Average of the Daily Morning Trough Peak Expiratory Flow (PEF) Over the 12 Week Treatment
Description: Morning PEF tests were performed before administration of study drug or rescue medications (data were excluded if the time of PEF measurement was more than 5 minutes after the dose time). The patient recorded the highest value of 3 measurements obtained in the patient diary.
  The baseline PEF was the average value of recorded (nonmissing) morning assessments over the 7 days prior to randomization on Day 1. For efficacy analyses of weekly average morning PEF measurements, values were the averages based on available data for that week.
Time Frame: Days -6 to Day 1 (predose, baseline), Day 1 (postdose) daily until Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: liters/minute
Arm/Group | FS MDPI 200 / 12.5 mcg | FS MDPI 100 / 12.5 mcg | Fp MDPI 200 mcg | Fp MDPI 100 mcg | Placebo MDPI
Number analyzed (Participants) | 145 | 141 | 146 | 145 | 142
liters/minute | 20.235 (2.3845) | 18.610 (2.4137) | 7.464 (2.3887) | 5.731 (2.4102) | -10.987 (2.4784)
Statistical Analysis 1: Comparison: Fp MDPI 200 mcg vs Placebo MDPI; The analysis of change from baseline in weekly average of daily (AM predose and pre rescue bronchodilator) PEF over the 12-week treatment period was performed using an mixed model for repeated measures (MMRM) with an unstructured covariance matrix and with effects due to baseline weekly average of daily AM PEF, sex, age, (pooled) center, previous therapy (ICS or ICS/LABA), week, treatment, and week-by-treatment interaction; Test type: Superiority or Other; p = 0.0000, mixed model for repeated measures — Significance level of 0.05; LSM difference = 18.450, 95% CI 2-sided [11.751 to 25.150]
Statistical Analysis 2: Comparison: Fp MDPI 100 mcg vs Placebo MDPI; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0000, mixed model for repeated measures — Significance level of 0.05; LSM difference = 16.718, 95% CI 2-sided [9.988 to 23.449]
Statistical Analysis 3: Comparison: FS MDPI 200 / 12.5 mcg vs Placebo MDPI; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0000, mixed model for repeated measures — Significance level of 0.05; LSM difference = 31.221, 95% CI 2-sided [24.513 to 37.930]
Statistical Analysis 4: Comparison: FS MDPI 100 / 12.5 mcg vs Placebo MDPI; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0000, mixed model for repeated measures — Significance level of 0.05; LSM difference = 29.597, 95% CI 2-sided [22.839 to 36.354]
Statistical Analysis 5: Comparison: FS MDPI 200 / 12.5 mcg vs Fp MDPI 200 mcg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0002, mixed model for repeated measures — Significance level of 0.05; LSM difference = 12.771, 95% CI 2-sided [6.179 to 19.363]
Statistical Analysis 6: Comparison: FS MDPI 100 / 12.5 mcg vs Fp MDPI 100 mcg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0002, mixed model for repeated measures — Significance level of 0.05; LSM difference = 12.879, 95% CI 2-sided [6.216 to 19.541]
Statistical Analysis 7: Comparison: FS MDPI 100 / 12.5 mcg vs Fp MDPI 200 mcg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0010, mixed model for repeated measures — Significance level of 0.05; LSM difference = 11.146, 95% CI 2-sided [4.511 to 17.782]

4. Secondary Outcome: Change From Baseline in the Weekly Average of the Total Daily Asthma Symptom Score Over the 12-Week Treatment Period
Description: The total daily asthma symptom score is the average of the daytime and nighttime scores as recorded in the patient diary.
  Daytime Symptom Score:
  * 0=No symptoms
  * 1=Symptoms for 1 short period
  * 2=Symptoms for 2+ short periods
  * 3=Symptoms for most of the day - did not affect normal daily activities
  * 4=Symptoms for most of the day - did affect normal daily activities
  * 5=Symptoms so severe that I could not go to work or perform normal daily activities
  Nighttime Symptom Score (determined in the AM):
  * 0=No symptoms
  * 1=Symptoms causing me to wake once (or wake early)
  * 2=Symptoms causing me to wake twice or more (including waking early)
  * 3=Symptoms causing me to be awake for most of the night
  * 4=Symptoms so severe that I did not sleep Baseline was the average of recorded scores over the 7 days before randomization. The change from baseline in the weekly average over weeks 1 to 12 was analyzed using an mixed model for repeated measures (MMRM).
Time Frame: Days -6 to Day 1 (predose, baseline), to Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | FS MDPI 200 / 12.5 mcg | FS MDPI 100 / 12.5 mcg | Fp MDPI 200 mcg | Fp MDPI 100 mcg | Placebo MDPI
Number analyzed (Participants) | 145 | 141 | 146 | 145 | 142
units on a scale | -0.391 (0.0328) | -0.364 (0.0332) | -0.242 (0.0329) | -0.282 (0.0333) | -0.087 (0.0342)
Statistical Analysis 1: Comparison: Fp MDPI 200 mcg vs Placebo MDPI; The change from baseline in the weekly average of the total daily asthma symptom scores over weeks 1 to 12 was analyzed using an MMRM with an unstructured covariance matrix and with effects due to baseline score, sex, age, (pooled) center, previous therapy (ICS or ICS/LABA), week, treatment, and week-by-treatment interaction; Test type: Superiority or Other; p = 0.0010, mixed model for repeated measures — Significance level of 0.05; LSM difference = -0.156, 95% CI 2-sided [-0.248 to -0.063]
Statistical Analysis 2: Comparison: Fp MDPI 100 mcg vs Placebo MDPI; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0000, mixed model for repeated measures — Significance level of 0.05; LSM difference = -0.195, 95% CI 2-sided [-0.288 to -0.102]
Statistical Analysis 3: Comparison: FS MDPI 200 / 12.5 mcg vs Placebo MDPI; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0000, mixed model for repeated measures — Significance level of 0.05; LSM difference = -0.304, 95% CI 2-sided [-0.397 to -0.212]
Statistical Analysis 4: Comparison: FS MDPI 100 / 12.5 mcg vs Placebo MDPI; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0000, mixed model for repeated measures — Significance level of 0.05; LSM difference = -0.277, 95% CI 2-sided [-0.370 to -0.184]
Statistical Analysis 5: Comparison: FS MDPI 200 / 12.5 mcg vs Fp MDPI 200 mcg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0014, mixed model for repeated measures — Significance level of 0.05; LSM difference = -0.149, 95% CI 2-sided [-0.239 to -0.058]
Statistical Analysis 6: Comparison: FS MDPI 100 / 12.5 mcg vs Fp MDPI 100 mcg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0818, mixed model for repeated measures — Significance level of 0.05; LSM difference = -0.082, 95% CI 2-sided [-0.174 to 0.010]
Statistical Analysis 7: Comparison: FS MDPI 100 / 12.5 mcg vs Fp MDPI 200 mcg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0094, mixed model for repeated measures — Significance level of 0.05; LSM difference = -0.121, 95% CI 2-sided [-0.213 to -0.030]

5. Secondary Outcome: Change From Baseline in the Weekly Average of the Total Daily (24-hour) Use of Albuterol/Salbutamol Inhalation Aerosol Over the 12-Week Treatment Period
Description: Patients recorded the number of inhalations of rescue medication (albuterol/salbutamol HFA MDI) each AM and PM in the diary. The average number of daily inhalations over the 7 days before the randomization visit was the baseline value. The weekly average was based on the available data for the 7 days before each analysis week.
  The change from baseline in the weekly average of total daily (24-hour) use of albuterol/ salbutamol inhalation aerosol (number of inhalations) over weeks 1 to 12 was analyzed using a mixed model for repeated measures.
Time Frame: Days -6 to Day 1 (predose, baseline), up to week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: puffs
Arm/Group | FS MDPI 200 / 12.5 mcg | FS MDPI 100 / 12.5 mcg | Fp MDPI 200 mcg | Fp MDPI 100 mcg | Placebo MDPI
Number analyzed (Participants) | 145 | 141 | 146 | 145 | 143
puffs | -0.898 (0.1069) | -0.821 (0.1080) | -0.534 (0.1070) | -0.439 (0.1081) | 0.168 (0.1102)
Statistical Analysis 1: Comparison: Fp MDPI 200 mcg vs Placebo MDPI; The change from baseline in the weekly average of total daily (24-hour) use of albuterol/ salbutamol inhalation aerosol (number of inhalations) over weeks 1 to 12 was analyzed using an MMRM with an unstructured covariance matrix and with effects due to baseline value, sex, age, (pooled) center, previous therapy (ICS or ICS/LABA), week, treatment, and week-by-treatment interaction; Test type: Superiority or Other; p = 0.0000, mixed model for repeated measures — Significance level of 0.05; LSM difference = -0.702, 95% CI 2-sided [-1.001 to -0.403]
Statistical Analysis 2: Comparison: Fp MDPI 100 mcg vs Placebo MDPI; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0001, mixed model for repeated measures — Significance level of 0.05; LSM difference = -0.607, 95% CI 2-sided [-0.908 to -0.307]
Statistical Analysis 3: Comparison: FS MDPI 200 / 12.5 mcg vs Placebo MDPI; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0000, mixed model for repeated measures — Significance level of 0.05; LSM difference = -1.066, 95% CI 2-sided [-1.365 to -0.766]
Statistical Analysis 4: Comparison: FS MDPI 100 / 12.5 mcg vs Placebo MDPI; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0000, mixed model for repeated measures — Significance level of 0.05; LSM difference = -0.989, 95% CI 2-sided [-1.291 to -0.686]
Statistical Analysis 5: Comparison: FS MDPI 200 / 12.5 mcg vs Fp MDPI 200 mcg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0160, mixed model for repeated measures — Significance level of 0.05; LSM difference = -0.364, 95% CI 2-sided [-0.659 to -0.068]
Statistical Analysis 6: Comparison: FS MDPI 100 / 12.5 mcg vs Fp MDPI 100 mcg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0124, mixed model for repeated measures — Significance level of 0.05; LSM difference = -0.382, 95% CI 2-sided [-0.681 to -0.083]
Statistical Analysis 7: Comparison: FS MDPI 100 / 12.5 mcg vs Fp MDPI 200 mcg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0588, Wilcoxon (Mann-Whitney) — Significance level of 0.05; LSM difference = -0.287, 95% CI 2-sided [-0.584 to 0.011]

6. Secondary Outcome: Kaplan-Meier Estimate of Probability of Remaining in Study At Week 12
Description: The analysis of probability of remaining in the study at Week 12 used the time to patient withdrawal for worsening asthma, defined as the number of days elapsed from the date of randomization to the date of withdrawal due to worsening asthma. Patients who were lost to follow-up, who had not withdrawn due to worsening asthma by week 12, or who had withdrawn due to reasons other than worsening asthma were right-censored at the date of last assessment.
Time Frame: up to Week 12 of the Treatment Period
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | FS MDPI 200 / 12.5 mcg | FS MDPI 100 / 12.5 mcg | Fp MDPI 200 mcg | Fp MDPI 100 mcg | Placebo MDPI
Number analyzed (Participants) | 145 | 141 | 146 | 145 | 143
probability | 0.9719 [0.927 to 0.989] | 0.9929 [0.950 to 0.999] | 0.9786 [0.935 to 0.993] | 0.9930 [0.951 to 0.999] | 0.8528 [0.781 to 0.903]
Statistical Analysis 1: Comparison: Fp MDPI 200 mcg vs Placebo MDPI; Test type: Superiority or Other; p = 0.0001, Log Rank — Significance level of 0.05
Statistical Analysis 2: Comparison: Fp MDPI 100 mcg vs Placebo MDPI; Test type: Superiority or Other; p < .0001, Log Rank — Significance level of 0.05
Statistical Analysis 3: Comparison: FS MDPI 200 / 12.5 mcg vs Placebo MDPI; Test type: Superiority or Other; p = 0.0003, Log Rank — Significance level of 0.05
Statistical Analysis 4: Comparison: FS MDPI 100 / 12.5 mcg vs Placebo MDPI; Test type: Superiority or Other; p < .0001, Log Rank — Significance level of 0.05
Statistical Analysis 5: Comparison: FS MDPI 200 / 12.5 mcg vs Fp MDPI 200 mcg; Test type: Superiority or Other; p = 0.7203, Log Rank — Significance level of 0.05
Statistical Analysis 6: Comparison: FS MDPI 100 / 12.5 mcg vs Fp MDPI 100 mcg; Test type: Superiority or Other; p = 0.9960, Log Rank — Significance level of 0.05
Statistical Analysis 7: Comparison: FS MDPI 100 / 12.5 mcg vs Fp MDPI 200 mcg; Test type: Superiority or Other; p = 0.3250, Log Rank — Significance level of 0.05

7. Secondary Outcome: Change From Baseline in the Asthma Quality of Life Questionnaire With Standardized Activities (AQLQ(S)) Score at Endpoint for Patients >=18 Years Old
Description: The AQLQ(S) (September 2010 version; patients aged ≥18 years) was self administered by the patients at the investigational center at the randomization visit and at Week 12 or end of trial. The questionnaire is a tool to measure the impact of asthma on a patient's quality of life (physical, emotional, social, and occupational) with a recall period of 2 weeks. The AQLQ(S) was administered only to patients 18 years and older. The 32 individual questions in the AQLQ were equally weighted. The overall AQLQ score was the mean of the responses to each of the 32 questions, and ranged from 1 to 7. A score 7.0 indicated that the patient had no impairments due to asthma and a score of 1.0 indicated severe impairment.
  Positive change from baseline scores indicate improved quality of life.
Time Frame: Day 1 (predose, baseline), end of trial (up to week 12)
Population: Full analysis set of participants who contributed at least once to analysis and were >= 18 years old
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | FS MDPI 200 / 12.5 mcg | FS MDPI 100 / 12.5 mcg | Fp MDPI 200 mcg | Fp MDPI 100 mcg | Placebo MDPI
Number analyzed (Participants) | 131 | 135 | 132 | 133 | 129
units on a scale | 0.534 (0.0741) | 0.592 (0.0725) | 0.384 (0.0742) | 0.340 (0.0740) | -0.089 (0.0747)
Statistical Analysis 1: Comparison: Fp MDPI 200 mcg vs Placebo MDPI; The change from baseline in AQLQ(S) score (patients ≥18 years of age) at endpoint (ie, last postbaseline observation) was analyzed using an ANCOVA model with effects due to baseline AQLQ(S) score, sex, age, (pooled) center, previous therapy (ICS or ICS/LABA), and treatment, imputing missing data via last observation carried forward (LOCF); Test type: Superiority or Other; p = 0.0000, ANCOVA — Significance level of 0.05; LSM difference = 0.473, 95% CI 2-sided [0.269 to 0.677]
Statistical Analysis 2: Comparison: Fp MDPI 100 mcg vs Placebo MDPI; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.0000, ANCOVA — Significance level of 0.05; LSM difference = 0.428, 95% CI 2-sided [0.224 to 0.632]
Statistical Analysis 3: Comparison: FS MDPI 200 / 12.5 mcg vs Placebo MDPI; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.0000, ANCOVA — Significance level of 0.05; LSM difference = 0.623, 95% CI 2-sided [0.418 to 0.828]
Statistical Analysis 4: Comparison: FS MDPI 100 / 12.5 mcg vs Placebo MDPI; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.0000, ANCOVA — Significance level of 0.05; Slope = 0.681, 95% CI 2-sided [0.478 to 0.885]
Statistical Analysis 5: Comparison: FS MDPI 200 / 12.5 mcg vs Fp MDPI 200 mcg; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.1490, ANCOVA — Significance level of 0.05; LSM difference = 0.150, 95% CI 2-sided [-0.054 to 0.354]
Statistical Analysis 6: Comparison: FS MDPI 100 / 12.5 mcg vs Fp MDPI 100 mcg; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.0143, ANCOVA — Significance level of 0.05; LSM difference = 0.253, 95% CI 2-sided [0.051 to 0.455]
Statistical Analysis 7: Comparison: FS MDPI 100 / 12.5 mcg vs Fp MDPI 200 mcg; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.0435, ANCOVA — Significance level of 0.05; LSM difference = 0.209, 95% CI 2-sided [0.006 to 0.411]

8. Secondary Outcome: Kaplan-Meier Estimates for Time to 15% and 12% Improvement From Baseline in FEV1 Postdose on Day 1
Description: The baseline forced expiratory volume in 1 second (FEV1) was the average of the 2 predose FEV1 measurements (30 and 10 minutes predose) on Day 1. If one of these was missing, the other measurement was used as baseline value. If both were missing, the baseline trough FEV1 was treated as missing.
  Time to target improvement (15% or 12%) was defined as the time elapsed from the time of first dose to the first time the target improvement in FEV1 was achieved. If an exact target increase was not achieved at a measured timepoint, then the time was estimated by linear interpolation between the timepoint when target was reached and the timepoint immediately before. Patients who did not achieve the target improvement were censored at the time of last serial spirometry assessment.
  Values of NA indicate the values could not be estimated which happened when the estimated probability of not achieving target is more than 50%.
Time Frame: Day 1 of the Treatment Period (predose and postdose)
Population: Patients who did not achieve the target improvement were censored at the time of last serial spirometry assessment.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | FS MDPI 200 / 12.5 mcg | FS MDPI 100 / 12.5 mcg | Fp MDPI 200 mcg | Fp MDPI 100 mcg | Placebo MDPI
Number analyzed (Participants) | 68 | 58 | 61 | 64 | 61
hours
  15% improvement | 0.8 [0.310 to 1.770] | 0.9 [0.480 to 11.960] | NA [3.840 to NA] — estimated probability of not achieving target is more than 50%. | NA [NA to NA] — estimated probability of not achieving target is more than 50%. | NA [NA to NA] — estimated probability of not achieving target is more than 50%.
  12% improvement | 0.4 [0.250 to 0.810] | 0.4 [0.290 to 1.680] | 6.9 [2.690 to NA] — estimated probability of not achieving target is more than 50%. | NA [5.580 to NA] — estimated probability of not achieving target is more than 50%. | NA [5.680 to NA] — estimated probability of not achieving target is more than 50%.

9. Secondary Outcome: Patients With Treatment-Emergent Adverse Experiences (TEAE) During the Treatment Period
Description: An adverse event was defined as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. Severity was rated by the investigator on a scale of mild, moderate and severe, with severe= an AE which prevents normal daily activities. Relation of AE to treatment was determined by the investigator. Serious AEs include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, OR an important medical event that jeopardized the patient and required medical intervention to prevent the previously listed serious outcomes.
Time Frame: Day 1 to Week 12 of the Treatment Period
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | FS MDPI 200 / 12.5 mcg | FS MDPI 100 / 12.5 mcg | Fp MDPI 200 mcg | Fp MDPI 100 mcg | Placebo MDPI
Number analyzed (Participants) | 145 | 143 | 146 | 145 | 144
Participants
  >=1 TEAE | 61 | 59 | 60 | 53 | 52
  >=1 severe TEAE | 3 | 2 | 0 | 1 | 1
  >=1 treatment-related TEAE | 8 | 4 | 9 | 6 | 5
  >=1 severe treatment-related TEAE | 1 | 0 | 0 | 0 | 0
  >=1 serious TEAE | 2 | 2 | 1 | 1 | 1
  >=1 TEAE leading to withdrawal | 2 | 2 | 0 | 2 | 2
  >=1 nonserious TEAE | 61 | 58 | 60 | 52 | 52
  >=1 TEAE resulting in death | 0 | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to Week 14
Groups:
- FS MDPI 100/12.5 mcg: Following randomization, participants in this treatment arm took 1 inhalation using a multidose dry powder inhaler (MDPI) twice a day of fluticasone propionate 100 mcg (for a total daily dose of 200 mcg) and salmeterol 12.5 mcg (for a total daily dose of 25 mcg) for 12 weeks.
  Albuterol/salmeterol HFA MDI: Albuterol/salmeterol hydrofluoroalkane (HFA) metered dose inhaler (MDI) was supplied to participants throughout the study to be used as needed as a rescue medication.
- FS MDPI 200/12.5 mcg: Following randomization, participants in this treatment arm took 1 inhalation twice a day using a multidose dry powder inhaler (MDPI) of fluticasone propionate 200 mcg (for a total daily dose of 400 mcg) and salmeterol 12.5 mcg (for a total daily dose of 25 mcg) for 12 weeks.
  Albuterol/salmeterol HFA MDI: Albuterol/salmeterol hydrofluoroalkane (HFA) metered dose inhaler (MDI) was supplied to participants throughout the study to be used as needed as a rescue medication.
- Placebo: Following randomization, participants in this treatment arm took 1 inhalation using a multidose dry powder inhaler (MDPI) twice a day of placebo for 12 weeks.
  Albuterol/salmeterol HFA MDI: Albuterol/salmeterol hydrofluoroalkane (HFA) metered dose inhaler (MDI) was supplied to participants throughout the study to be used as needed as a rescue medication.
Arm/Group | FS MDPI 100/12.5 mcg | FS MDPI 200/12.5 mcg | Fp MDPI 100 mcg | Fp MDPI 200 mcg | Placebo
Serious Adverse Events (participants affected / at risk) | 2/143 | 2/145 | 1/145 | 1/146 | 1/144
Other Adverse Events (participants affected / at risk) | 21/143 | 20/145 | 26/145 | 20/146 | 20/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FS MDPI 100/12.5 mcg (N=143) | FS MDPI 200/12.5 mcg (N=145) | Fp MDPI 100 mcg (N=145) | Fp MDPI 200 mcg (N=146) | Placebo (N=144)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Grand mal convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FS MDPI 100/12.5 mcg (N=143) | FS MDPI 200/12.5 mcg (N=145) | Fp MDPI 100 mcg (N=145) | Fp MDPI 200 mcg (N=146) | Placebo (N=144)
Nasopharyngitis (Infections and infestations) | 10 (10) | 10 (12) | 7 (7) | 7 (8) | 8 (9)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 6 (6) | 9 (11) | 8 (9) | 7 (7)
Headache (Nervous system disorders) | 6 (21) | 4 (5) | 11 (18) | 7 (7) | 7 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.